CLINICAL TRIAL: NCT05780476
Title: A Novel Virtual Reality Intervention for Caregivers of People With Dementia.
Brief Title: A Novel VIRTUAL Reality Intervention for CAREgivers of People With Dementia (VirtualCare)
Acronym: VirtualCare
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: IRCCS Centro San Giovanni di Dio Fatebenefratelli (Other)
Collaborators: Alzheimer's Association (Other); University of Bergamo (Other)
Responsible Party: Principal Investigator, Cristina Festari, PhD, Researcher, IRCCS Centro San Giovanni di Dio Fatebenefratelli
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: AACSF-22-924470
Record Dates: First submitted 2023-02-28; First posted 2023-03-22 (Actual); Last update posted 2023-03-22 (Actual); Status verified 2023-03

CONDITIONS: Caregiver Burden
Keywords: Informal caregiver; Virtual reality; Psychoeducation intervention
MeSH Terms: conditions — Caregiver Burden

STUDY DESIGN:
Intervention Model Description: Two-arm randomized controlled design
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Active Comparator): Psychoeducational program.
  Interventions: Behavioral: Psychoeducation
- Experimental group (Experimental): Psychoeducational program combined with virtual reality.
  Interventions: Behavioral: Psychoeducation + virtual reality

INTERVENTIONS:
Behavioral: Psychoeducation — 6 sessions of 2 hours over 6 weeks
  Arms: Control group
Behavioral: Psychoeducation + virtual reality — 6 sessions of 2 hours over 6 weeks. Virtual reality experience will be carry out in the last 30 minutes of each meeting. Virtual reality consists of 360-degree videos depicting everyday situations and allowing the caregivers to feel the specific symptoms of dementia (e.g., disorientation, agnosia, apraxia and memory loss).
  Arms: Experimental group

SUMMARY:
This clinical trial aims to explore if a virtual reality experience increases the beneficial effect of psychoeducational programs in informal caregivers of people with mild-to-moderate Alzheimer's disease. This study will test changes in psychological distress and neural activity in brain systems that regulate stress and empathic care.

Participants will be randomized into two arms: the control group will participate in an online psychoeducational intervention, while the experimental group will participate in the psychoeducational intervention combined with virtual reality.

ELIGIBILITY:
Inclusion Criteria:

* Being an unpaid informal caregiver (CG; i.e., family members or friends) living with or caring for a person with Alzheimer's Disease (AD) for at least 4 hours a day for at least six months before enrolment;
* Caring for a person with a diagnosis of AD at prodromal or mild stage (i.e., Mini-Mental State Examination score:18-24) and still living at home.

Exclusion Criteria:

* Receiving daily assistance for more than 10 hours from formal CGs;
* Being formal CGs (i.e., nurse or another paid figure);
* Being informal CGs of i) persons with moderate-to-severe AD, or ii) persons with non-AD diseases;
* Not having or being able to use a device connected to internet (e.g., smartphones or PC).
* Having received psychotherapeutic o psychological support, or having already participated to psychoeducational programs.
* Only a family member for person with dementia is accepted.

Exclusion Criteria for experimental group (Psychoeducation + VR):

* Medical history of epilepsy.

Exclusion Criteria for subsample of caregivers assess with MRI:

* Metal implants, artificial prostheses, pace-makers, prosthetic heart valves;
* Claustrophobia;
* Pregnancy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in distress of care after intervention | Baseline (pre-intervention); Post-intervention (up to a week post-intervention).
  Zarit Burden interview - ZBI
Change in anxiety | Baseline (pre-intervention); Post-intervention (up to a week post-intervention).
  State Trait Anxiety Inventory - STAI-Y

SECONDARY OUTCOMES:
Change in empathy | Baseline (pre-intervention); Post-intervention (up to a week post-intervention).
  Interpersonal Reactivity Index - IRI
Change in sense of competence | Baseline (pre-intervention); Post-intervention (up to a week post-intervention).
  Short sense of competence questionnaire - SSCQ
Modulation of neural activity in brain systems regulating empathy | Baseline (pre-intervention); Post-intervention (up to a week post-intervention).
  Task fMRI

OTHER OUTCOMES:
Persistence of medium-term effects - distress of care | 2 months post-intervention.
  Zarit Burden interview - ZBI
Persistence of medium-term effects - anxiety | 2 months post-intervention.
  State Trait Anxiety Inventory - STAI-Y
Persistence of medium-term effects - empathy | 2 months post-intervention.
  Interpersonal Reactivity Index - IRI
Persistence of medium-term effects - sense of competence | 2 months post-intervention.
  Short sense of competence questionnaire - SSCQ

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Festari, PhD, Principal Investigator — IRCCS Istituto Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy
Locations (1):
- IRCCS Centro San Giovanni di Dio Fatebenefratelli, Brescia, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Morganti F, Palena N, Savoldelli P, Greco A. Take the First-Person Perspective to Become Dementia-Friendly: The Use of 360 degrees Video for Experiencing Everyday-Life Challenges With Cognitive Decline. Front Psychol. 2020 Jun 30;11:1117. doi: 10.3389/fpsyg.2020.01117. eCollection 2020. PMID 32695039
- [Derived] Singh Solorzano C, Bonomini C, Rosini S, Passeggia I, Zanetti O, Pievani M, Frisoni GB, Festari C. The psychological impact of the disclosure of the diagnosis of Alzheimer's disease on informal caregivers. Alzheimers Dement. 2025 Sep;21(9):e70412. doi: 10.1002/alz.70412. PMID 40908671
- [Derived] Festari C, Bonomini C, Rosini S, Gattuso M, Singh Solorzano C, Zanetti O, Corbo D, Agnelli G, Quattrini G, Ferrari C, Gasparotti R, Pievani M, Morganti F. Virtual Reality Combined With Psychoeducation to Improve Emotional Well-Being in Informal Caregivers of Alzheimer's Disease Patients: Rationale and Study Design of a Randomized Controlled Trial. Int J Geriatr Psychiatry. 2024 Sep;39(9):e6145. doi: 10.1002/gps.6145. PMID 39267224